CLINICAL TRIAL: NCT02925286
Title: Effects of a Workplace Prevention Program for Problematic Gambling
Acronym: Alna
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stockholm University (Other)
Collaborators: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Per Carlbring, Professor, Stockholm University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Alna
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Gambling
Keywords: gambling prevention; workplace policy
MeSH Terms: conditions — Gambling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Five organizations will get the intervention during fall/winter 2016.
  Interventions: Other: Prevention program for gambling in the workplace
- Wait-list group (No Intervention): Five organizations will be on the waitlist for 12 months and then get the intervention.

INTERVENTIONS:
Other: Prevention program for gambling in the workplace — The intervention group will receive a gambling prevention program which includes generating and implementing policies and education on addiction and gambling. The full length of the program will be about 14 hours.
  Arms: Intervention group

SUMMARY:
The purpose of this study is to determine the effects of a workplace prevention program targeting problematic gambling.

DETAILED DESCRIPTION:
There is a considerable knowledge-gap regarding the efficacy of problem gambling prevention in workplace settings. At the same time, this knowledge is widely requested upon both by researchers and government agencies. The evaluation of prevention programs is important both in a public health perspective and for the organizations investing in preventive interventions for problem gambling at the workspaces and the current study aims to contribute with knowledge regarding the potential effects of such an intervention.

The purpose of this study is to determine the effects of a workplace prevention program regarding problematic gambling, on a variety of outcomes. The authors hypothesize that the program will lead to differences in:

* A change in gambling habits among coworkers and managers
* That fewer workers and managers will report problem gambling
* That the managers who participate in the intervention will report being more confident in handling gambling and problem gambling at the workplace
* That the managers who participate in the intervention will report a higher inclination to engage in a conversation with an employee when suspicion or worry about problem gambling arises
* That the number of actions to help employees with problem gambling or other types of harmful use will raise among organizations who participate in the intervention.
* An increase in the employees' knowledge about what kind of support regarding gambling or addiction is available from the workplace and where to find it.

ELIGIBILITY:
Program Inclusion Criteria:

* To be eligible to participate in the workplace program, the participant must be currently employed as manager in one of the organizations that will participate in the study

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5625 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2017-11-30 (Actual)

PRIMARY OUTCOMES:
Survey question about supervisors perceived inclination to initiate a conversation with an employee when worry or suspicion of problematic gambling or other harmful use arises. | Change from baseline at: [1] 3 months after baseline, [2] 12 months after baseline, and [3] 24 months past baseline.

SECONDARY OUTCOMES:
Survey questions about supervisors and workers gambling frequencies | [1] 3 months after baseline (Supervisors only) , [2] 12 months after baseline, and [3] 24 months past baseline.
  Gambling frequencies online/offline in the last 1 and 12 month(s).
Survey questions about knowledge of present policies and where to go for help | [1] 3 months after baseline (Supervisors only) , [2] 12 months after baseline, and [3] 24 months past baseline.
Survey questions regarding worrying about, or acting to help, co-workers | [1] 3 months after baseline (Supervisors only) , [2] 12 months after baseline, and [3] 24 months past baseline.
Survey question regarding knowledge about whether co-workers gamble during work | [1] 3 months after baseline (Supervisors only) , [2] 12 months after baseline, and [3] 24 months past baseline.
The Problem Gambling Severity Index (PGSI) | [1] 3 months after baseline (Supervisors only) , [2] 12 months after baseline, and [3] 24 months past baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Per Carlbring, Professor, Principal Investigator — Stockholm University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rafi J, Ivanova E, Rozental A, Carlbring P. Effects of a workplace prevention programme for problem gambling: study protocol for a cluster randomised controlled trial. BMJ Open. 2017 Sep 25;7(9):e015963. doi: 10.1136/bmjopen-2017-015963. PMID 28951403